CLINICAL TRIAL: NCT00479622
Title: A Randomized, Two-Arm, Parallel Group Study of the Safety, Pharmacokinetics, and Pharmacodynamics of TRU-015 Added to Standard Therapy in Subjects With Membranous Nephropathy Secondary to Systemic Lupus Erythematosus
Brief Title: Study of TRU-015 in Subjects With Membranous Nephropathy Secondary to Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Emergent Product Development Seattle LLC (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3206K3-103
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Membranous Nephropathy; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Glomerulonephritis, Membranous | interventions — TRU-015 protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: TRU-015
- 2 (Experimental)
  Interventions: Drug: TRU-015

INTERVENTIONS:
Drug: TRU-015 — Arm 1 = 800 mg Arm 2 = 2000 mg

SUMMARY:
The purpose of this study is to determine how the body absorbs and chemically changes a single infusion of TRU-015 in subjects with kidney disease caused by lupus.

ELIGIBILITY:
Inclusion Criteria:

* Man or nonlactating and nonpregnant woman, aged 18 to 70 years, inclusive, at the screening visit.
* Diagnosis of systemic lupus erythematosus more than 6 months before study day 1.
* History of positive antinuclear antibody titer of >1:160 or equivalent.
* Biopsy-proven class V lupus nephritis within the last 2 years.
* Have been on a stable dose of oral corticosteroids (<20 mg/day prednisone or equivalent) for 2 months before study day 1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of TRU-015 after a single administration in subjects with membranous nephropathy secondary to systemic lupus erythematosus. | 6 months

SECONDARY OUTCOMES:
To evaluate the safety, immunogenicity, and pharmacokinetic/pharmacodynamic relationship of TRU-015 in subjects with membranous nephropathy secondary to systemic lupus erythematosus. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (6):
- United States (6):
  - Los Angeles, California
  - Palo Alto, California
  - Lake Success, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Columbus, Ohio